CLINICAL TRIAL: NCT04425759
Title: Prevalence and Risk Factors of SARS-CoV-2 Antibody Responses and Assymptomatic Carriers Among a Cohort of 2,300 Healthcare Workers at the Consorci Sanitari Del Maresme (CSdM)
Brief Title: Prevalence and Risk Factors of SARS-CoV-2 Antibody Responses (COVID-19)
Acronym: SERO-MARES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, Director of Research and Academic Development at CSdM, Hospital de Mataró
Other Study IDs: SERO-MARES (56/20)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Covid19; Corona Virus Infection; SARS-CoV 2; COVID
Keywords: COVID; ANTIBODY; SARS-COV2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood sammples for the serological analysis will be collected at 0/90/180/270/360 days.

SUMMARY:
Observational and prospective study with one year of follow-up of the cohort of workers of the CSdM, including workers of subcontracted companies working in the Hospital of Mataró (2,300 workers approximately) and with controls at baseline and at 3, 6, 9 and 12 months. All CSdM workers will be invited to participate by e-mail and by announcements in the corporate website. A space will be set up on the corporate intranet where workers will be informed about the study, will be able to give their informed consent and will be able to answer an electronic questionnaire regarding socio-demographic, clinical and labour personal characteristics. Once the questionnaire answered, participants will be authorized to schedule a blood extraction. Prevalence of antibodies against SARS-CoV-2 will be analyzed (IgA, IgM, IgG). PCR will be also performed for IgM and IgA positive subjects.

DETAILED DESCRIPTION:
* Study design: observational and prospective study with one year of follow-up of the cohort of workers of the CSdM, including workers of subcontracted companies working in the Hospital of Mataró (2,300 workers approximately) and with controls at baseline and at 3, 6, 9 and 12 months.
* Aims: to perform a universal test for all the professionals of the Consorci Sanitari del Maresme (CSdM) in order to carry out the following objectives:

  1. Let them know if they have been exposed to the SARS-CoV-2 virus.
  2. Identify asymptomatic carriers of SARS-CoV-2 virus.
  3. Develop an immune map of all the professionals to: a) describe the seroprevalence of SARS-CoV-2 antibodies and their evolution over a year; b) help minimize the risk of infection in CSdM professionals; c) contribute to the improvement of knowledge about the infection and the social and occupational factors that affect its spread; and d) allow in the future to identify the duration of immunity against SARS-CoV-2.
* Time Frame: 1 year.
* Study population: all workers from the healthcare centers of the Consorci Sanitari del Maresme will be invited to participate by e-mail and by announcements in the corporate website. A space will be set up on the corporate intranet where workers will be informed about the study, will be able to give their informed consent and will be able to answer an electronic questionnaire regarding socio-demographic, clinical and labour personal characteristics. Once the questionnaire answered, participants will be authorized to schedule a blood extraction.
* Methods: Prevalence of antibodies against SARS-CoV-2 will be analyzed (IgA, IgM, IgG) and PCR will be also performed for IgM and IgA positive subjects following this algorithm:

Serological study:

1. Screening the entire population with total CLIA result (IgA, IgM, IgG) to determine negatives.
2. ELISA for positives with differentiated IgM, IgA and IgG results.
3. PCR of nasopharyngeal smears on all IgM and IgA + (to determine asymptomatic cases).

There will be other blood samplings and determination points at 3, 6, 9 and 12 months for all the study participants.

ELIGIBILITY:
Inclusion Criteria:

* All the professionals working at the Consorci Sanitari del Maresme (approximately 2300 subjects).

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professionals working at the Maresme Health Consortium (CSdM).
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Antibodies to SARS-CoV2: IgA, IgM, IgG | 1 year
  * Screening for the entire population with total IgA, IgM, IgG to screen the negatives
  * ELISA for positives with differentiated IgM+IgA vs IgG specific for SARS-Cov-2 seroprevalence of SARS-CoV-2 antibodies and their evolution over a year; b) help minimize the risk of infection in CSdM professionals; c) contribute to the improvement of knowledge about the infection and the social and occupational factors that affect its spread; and d) allow in the future to identify the duration of immunity against SARS-CoV-2.
PCR of nasopharyngeal smears on all IgM + | 1 year
  * To detect symptomatic or asymptomatic carriers
  * New diagnostics of COVID19 confirmed by PCR of nasopharyngeal smears

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, MD, PhD, Principal Investigator — Hospital de Mataró
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No